CLINICAL TRIAL: NCT02354820
Title: Child Health Improvement Through Computer Automation of Constipation Management in Primary Care
Acronym: CHICA-GI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William E. Bennett, Jr. (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, William E. Bennett, Jr., Assistant Professor of Pediatrics, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHICA-GI Constipation; K23DK098235 (NIH)
Record Dates: First submitted 2015-01-26; First posted 2015-02-03 (Estimated); Results first posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Constipation; Encopresis
MeSH Terms: conditions — Constipation; Encopresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients are identified by the pre-screener form given to parents as having constipation or encopresis. No intervention is given to providers to help them with constipation management.
- Experimental (Experimental): Patients are identified by the pre-screener form given to parents as having constipation or encopresis. Evidence based reminders and patient educational materials are given to providers to help them with constipation management.
  Interventions: Other: Evidence Based Constipation Reminders

INTERVENTIONS:
Other: Evidence Based Constipation Reminders
  Arms: Experimental

SUMMARY:
This project seeks to expand an existing computerized decision support system used in pediatric primary care. The expanded system will add a module that helps clinicians recognize constipated children and then provides evidence-based reminders for constipation management, as well as automates patient educational materials. The current system is deployed across multiple sites, and the constipation module will be randomized to deployment in different sites. The difference in constipation management and patient outcomes will then be compared between sites receiving the intervention and sites not receiving the intervention over a 12 month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to one of 5 primary care clinics in the Eskenazi Health system in Indianapolis, IN.
* Patients given a pre-screener form as part of the existing CHICA decision support system.
* Age between 2 years and 12 years, inclusive.

Exclusion Criteria:

* None.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16264 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Patients are identified by the pre-screener form given to parents as having constipation or encopresis. Evidence based reminders and patient educational materials are given to providers to help them with constipation management.
  Evidence Based Constipation Reminders
Period: Overall Study
Arm/Group | Control | Experimental
Started | 9667 | 6597
Completed | 9667 | 6597
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 9667 | 6597 | 16264
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9667 | 6597 | 16264
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6 [3 to 9] | 6 [3 to 9] | 6 [3 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4752 | 3283 | 8035
  Male | 4915 | 3314 | 8229
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4431 | 3447 | 7878
  White | 907 | 683 | 1590
  More than one race | 4329 | 2467 | 6796
  Unknown or Not Reported | 0 | 0 | 0
Symptoms of constipation [Number; unit: participants] | 612 | 432 | 1044

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Persistent Constipation Within 6 Months
Description: Parents are asked if constipation is still present at a subsequent visit within 6 months.
Time Frame: All visits within 6 months of initial constipation complaint.
Measure: Number; unit: participants with persistent symptoms
Arm/Group | Control | Experimental
Number analyzed (Participants) | 4324 | 3153
participants with persistent symptoms | 325 | 224

ADVERSE EVENTS:
Arm/Group | Control | Experimental
Serious Adverse Events (participants affected / at risk) | 0/9667 | 0/6597
Other Adverse Events (participants affected / at risk) | 0/9667 | 0/6597

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes